CLINICAL TRIAL: NCT02169908
Title: LIPIDOXA, a Pilot Study of Analysis of Chronic Neuropathic Pain Markers in Patients Treated With Oxaliplatin-based Regimen
Brief Title: Analysis of Chronic Neuropathic Pain Markers in Patients Treated With Oxaliplatin
Acronym: LIPIDOXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LIPIDOXA
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Digestive Cancer; Gynecological Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

ARMS (1):
- Occurrence of painful neuropathy (Other): Assessment of neuropathic pain with two devices (Thermotest and von Frey hairs) and with the Neuropathic Pain Symptom Inventory.
  Interventions: Device: Thermotest; Device: von Frey hairs

INTERVENTIONS:
Device: Thermotest
Device: von Frey hairs

SUMMARY:
The role of oxidative stress in the development of oxaliplatin-induced peripheral neuropathy has been previously described in mice and in neuronal cell cultures (Massicot 2013); clinical manifestations and pathophysiological mechanisms potentially involved have also been described in humans (Andreas 2007) (Attal 2009).

The investigators team plans to conduct a translational clinicobiological research to explain the nature of the biochemical and molecular mechanisms of the development of oxaliplatin-induced painful neuropathy. To perform this project, the investigators propose to realize a pilot study in patients newly treated with oxaliplatin. This will be conducted in the oncology department of Paris Saint Joseph Hospital from May 2014 until the inclusion of 20 patients.

The main objective of this pilot study is to evaluate the occurrence of acute and chronic neuropathic pain occurring in patients newly treated with oxaliplatin. The characterization of this pain is based on validated tests (Cruccu 2010).

Moreover, the biochemical changes related to oxidative stress and those related to cellular lipid composition are characterized in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly traeted with oxaliplatin
* Patient suffering from any type of cancer treated with oxaliplatin
* Man or Woman over 18

Exclusion Criteria:

* Patient with brain or leptomeningeal metastases
* Patient previously treated with cisplatin
* Patient addicted to alcohol
* Diabetic patient with peripheral neurological disorders
* Patient receiving calcium or magnesium salts intravenously
* Patient suffering from peripheral neuropathy
* Patient suffering from psychiatric disorders
* Patient treated with at least one of the following drug: venlafaxine, carbamazepine, gabapentin, pregabalin, clomipramine, amitriptyline, imipramine, duloxetine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Thermal thresholds | Three to six months
  Four thermal thresholds are assessed by a Thermotest (Somedic AB):
  * cold perception threshold
  * warm perception threshold
  * cold pain threshold
  * warm pain threshold

SECONDARY OUTCOMES:
Tactile sensitivity | Three to six months
  Tactile sensitivity is assessed with von Frey hairs.

OTHER OUTCOMES:
Characterization of pain neuropathy | Three to six months
  Neuropathic Pain Symptom Inventory (NPSI questionnaire) is used.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Massicot F, Hache G, David L, Chen D, Leuxe C, Garnier-Legrand L, Rat P, Laprevote O, Coudore F. P2X7 Cell Death Receptor Activation and Mitochondrial Impairment in Oxaliplatin-Induced Apoptosis and Neuronal Injury: Cellular Mechanisms and In Vivo Approach. PLoS One. 2013 Jun 27;8(6):e66830. doi: 10.1371/journal.pone.0066830. Print 2013. PMID 23826152
- [Background] Binder A, Stengel M, Maag R, Wasner G, Schoch R, Moosig F, Schommer B, Baron R. Pain in oxaliplatin-induced neuropathy--sensitisation in the peripheral and central nociceptive system. Eur J Cancer. 2007 Dec;43(18):2658-63. doi: 10.1016/j.ejca.2007.07.030. Epub 2007 Sep 12. PMID 17855072
- [Background] Attal N, Bouhassira D, Gautron M, Vaillant JN, Mitry E, Lepere C, Rougier P, Guirimand F. Thermal hyperalgesia as a marker of oxaliplatin neurotoxicity: a prospective quantified sensory assessment study. Pain. 2009 Aug;144(3):245-252. doi: 10.1016/j.pain.2009.03.024. Epub 2009 May 19. PMID 19457614
- [Background] Cruccu G, Sommer C, Anand P, Attal N, Baron R, Garcia-Larrea L, Haanpaa M, Jensen TS, Serra J, Treede RD. EFNS guidelines on neuropathic pain assessment: revised 2009. Eur J Neurol. 2010 Aug;17(8):1010-8. doi: 10.1111/j.1468-1331.2010.02969.x. Epub 2010 Mar 8. PMID 20298428